CLINICAL TRIAL: NCT05226585
Title: Mechanisms of Change in Cognitive Behavioral Therapy for Insomnia (CBTi): A Randomized Controlled Pilot Trial
Brief Title: Mechanisms of Change in Cognitive Behavioral Therapy for Insomnia (CBTi)
Acronym: CBTi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2107024013
Record Dates: First submitted 2021-09-28; First posted 2022-02-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: insomnia; insomnia disorder; cognitive behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Three treatment arms and a waitlist control
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will not be aware of participant study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- In-person CBTi (Active Comparator): CBTi of variable treatment length will be administered by trained study staff in-person.
  Interventions: Behavioral: In-Person Cognitive Behavioral Therapy for Insomnia
- Telehealth CBTi (Active Comparator): CBTi of variable treatment length will be administered by trained study staff via HIPAA-compliant tele-video conference.
  Interventions: Behavioral: Telehealth Cognitive Behavioral Therapy for Insomnia
- Internet CBTi (Active Comparator): Self-paced CBTi of variable treatment length will be administered via Sleep Healthy Using The Internet (SHUTi).
  Interventions: Behavioral: Internet Cognitive Behavioral Therapy for Insomnia
- Waitlist Control (No Intervention): Treatment will be postponed by 12 weeks.

INTERVENTIONS:
Behavioral: In-Person Cognitive Behavioral Therapy for Insomnia — Cognitive behavioral therapy is recommended as a first-line treatment for insomnia (CBTi). CBTi contains the following well-validated components of cognitive behavioral treatment for insomnia: stimulus control, sleep compression, sleep hygiene, relaxation training, and cognitive restructuring.
  Other Names: CBTi
  Arms: In-person CBTi
Behavioral: Telehealth Cognitive Behavioral Therapy for Insomnia — Telehealth cognitive behavioral therapy is recommended as a first-line treatment for insomnia (CBTi) conducted via audio-video communication. tCBTi contains the following well-validated components of cognitive-behavioral treatment for insomnia: stimulus control, sleep compression, sleep hygiene, relaxation training, and cognitive restructuring.
  Other Names: tCBTi
  Arms: Telehealth CBTi
Behavioral: Internet Cognitive Behavioral Therapy for Insomnia — Sleep Healthy Using The Internet (SHUTi; aka iCBTi) is a self-guided, fully automated, online CBTi program that includes interactive features: personalized goal setting, graphical feedback based on inputted data, animations/illustrations to enhance comprehension, patient vignettes, and video-based expert explanations.
  Other Names: iCBTi
  Arms: Internet CBTi

SUMMARY:
The purpose of this study is to investigate the mechanisms of change in Cognitive Behavioral Therapy for insomnia (CBTi) in a sample of adults aged 50-65. This study aims to evaluate the pre-post treatment change in sleep, circadian rhythms, biomarkers, cognitive performance, and structural and functional magnetic resonance imaging scans (MRI).

DETAILED DESCRIPTION:
Baseline Part 1:

* Online demographic and contact information
* Schedule Baseline Part 2 with the investigators via online link
* 1 week of daily sleep diaries

Baseline Part 2:

* Internet-based interview with the investigators to confirm study eligibility requirements
* Online self-report questionnaires
* 2 weeks of daily sleep diaries
* 2 weeks of sleep/wake assessment wearing a watch-like activity monitor (Actiwatch)

Objective Baseline:

* Single-night, diagnostic in-home sleep study, including and the following equipment:

  * Adhesive patch which will adhere to the arm
  * Sensor belts worn around the chest, fitted with nasal canula, pulse oximeter, and 3 electrodes which will adhere to the back of the neck and behind each ear
* Next-day appointment:

  * Neuropsychological assessment
  * Structural and functional magnetic resonance imaging scan (MRI)
  * Non-invasive blood pressure readings
  * Low-volume Blood draw (used to obtain genetic biomarkers)
  * Removal of adhesive patch
* Next-day evening (2-nights):

  * Consumable capsule
  * Sensor belt worn around the chest/abdomen Random Assignment: If it is determined the participant is eligible for the study, participants will be randomly assigned to one of the treatment groups (in-person, telehealth or internet delivered) or asked to wait to start treatment.

Treatment Phase I:

* Participants will complete up to 12 weeks of insomnia treatment or wait for treatment ("waitlist") 12-Week Post-treatment Part 1:
* Complete 2 weeks of an online daily sleep diary and actigraphy
* Complete online self-report questionnaires

Objective 12-Week Post-treatment:

• Repeat "Objective Baseline" outlined above

Treatment Phase II (WLC):

* Treatment will start for participants who had been assigned to the waitlist condition 3-Month Follow-Up:
* Complete online self-report questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-65
* Normal hearing with or without hearing aids
* Ability to speak and read English and ability to give informed consent
* Possession of a computer with video and audio capabilities
* Meets DSM-5 Criteria for Insomnia Disorder
* Internet speed sufficient for participating in teletherapy (e.g., Zoom Health) or SHUTi (for iCBTi group)
* MoCA scores ≥24 will be deemed normal cognitive status and considered eligible for study participation and/or assessed by the ability to comprehend the baseline screening questionnaires
* Willing to refrain from new external behavioral health or medication treatment for issues pertaining to sleep during participation in the study
* Indication that the individual plans to be in the area for the 6 months following the first baseline assessment

Exclusion Criteria:

* Failure to meet the above "inclusion criteria"
* Current circadian rhythm disorder, sleep deprivation, or hypersomnia and related sleep disorders (assessed with clinical interview and/or self-report) as CBTi has not been validated in these populations. Verified by self-report and/or clinical interview (SCISD-R)
* Untreated sleep disordered breathing (e.g., obstructive sleep apnea) assessed by self-report, clinical interview, and/or diagnostic sleep study (i.e., baseline sleep study PSG)
* Failing to meet criteria for MRI scan (e.g., having metallic implants); see Pre-screen MRI Checklist for full list of exclusions for MRI scans.
* Fear/phobia of needles (conflict with blood draw) and/or small spaces (conflict with MRI scanner)
* Current suicide risk meriting crisis intervention as assessed by the Patient Health Questionnaire (PHQ-9) and/or disclosure of serious suicidal ideation
* Pregnancy (self-report, proposed instruments and treatments have not been validated in this population)
* Sleep efficiency > 85%, assessed by the sleep diary
* Serious mental health diagnosis (e.g., bipolar disorder or psychosis) assessed by structured interview (M.I.N.I.)
* Currently engaged in evidence-based psychotherapy for Insomnia (i.e., Cognitive Behavioral Therapy) by self-report
* Failure to follow protocol (e.g., consistent "no show" for appointments, answering questionnaires dishonestly, refusal to complete more than 2 assessments [e.g., fMRI and Neuropsych])

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Pre-treatment
  Self-reported severity of insomnia symptoms is assessed once at baseline.
Insomnia Severity Index | During treatment
  Self-reported severity of insomnia symptoms is assessed weekly through the duration of treatment.
Insomnia Severity Index | 12-week Post-treatment
  Self-reported severity of insomnia symptoms is assessed once at posttreatment.

SECONDARY OUTCOMES:
Diary-assessed Sleep | Pre-treatment
  Self-reported severity of sleep parameters (e.g., sleep efficiency, total sleep time, total time in bed).
Diary-assessed Sleep | During treatment
  Self-reported severity of sleep parameters (e.g., sleep efficiency, total sleep time, total time in bed).
Diary-assessed Sleep | 12 week Post-treatment
  Self-reported severity of sleep parameters (e.g., sleep efficiency, total sleep time, total time in bed).

OTHER OUTCOMES:
Circadian Rhythm | Pre-treatment
  Circadian rhythms as assessed by core body temperature
Circadian Rhythm | 12 week Post-treatment
  Circadian rhythms as assessed by core body temperature
Magnetic resonance imaging (MRI) | Pre-treatment
  Neurological outcomes (e.g., MRI resting-state functional connectivity: cingulate cortex, left insula, left cuneus, and fusiform; salience, executive control, and default mode networks.)
Magnetic resonance imaging (MRI) | 12 week Post-treatment
  Neurological outcomes (e.g., MRI resting-state functional connectivity: cingulate cortex, left insula, left cuneus, and fusiform; salience, executive control, and default mode networks.)
Inflammatory Health | 12 week Pre-treatment
  Cytokines (e.g., IL-6, IL-10, TNFalpha, GFAP, Tau, NFL, UCHL1)
Inflammatory Health | 12 week Post-treatment
  Cytokines (e.g., IL-6, IL-10, TNFalpha, GFAP, Tau, NFL, UCHL1)
Evaluation of executive functioning | Pre-treatment
  Neuropsychological tests of executive functioning using a program administered via iPad
Evaluation of episodic memory | Pre-treatment
  Neuropsychological tests of episodic memory using a program administered via iPad
Evaluation of executive functioning | 12 week Post-treatment
  Neuropsychological tests of executive functioning using a program administered via iPad. Due to the nature of these assessments, specific details of the tests cannot be disclosed.
Evaluation of episodic memory | 12 week Post-treatment
  Neuropsychological tests of episodic memory using a program administered via iPad. Due to the nature of these assessments, specific details of the tests cannot be disclosed.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Taylor, Ph.D., Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No